CLINICAL TRIAL: NCT02698527
Title: The Effect of Buffered Lidocaine Versus Nonbuffered Lidocaine on Pain Scores During Infiltration for Vulvar Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Jennifer C Villavicencio, Principal Invesitgator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14-0130
Record Dates: First submitted 2015-05-18; First posted 2016-03-03 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Genital Diseases, Female
Keywords: lidocaine
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Buffered Lidocaine (Active Comparator): Vulvar biopsy conducted using non-buffered lidocaine as anesthesia
  Interventions: Drug: Non-Buffered Lidocaine
- Buffered Lidocaine (Experimental): Vulvar biopsy conducted using buffered lidocaine as anesthesia
  Interventions: Drug: Buffered Lidocaine

INTERVENTIONS:
Drug: Non-Buffered Lidocaine — Active comparator
  Arms: Non-Buffered Lidocaine
Drug: Buffered Lidocaine — Experimental, additIon of Sodium Bicarbonate to Lidocaine
  Arms: Buffered Lidocaine

SUMMARY:
Objective: To compare pain scores on a visual analogue scale during infiltration of local anesthetic for vulvar biopsies between women who are treated with buffered versus non- buffered lidocaine

Hypothesis: Patients treated with buffered lidocaine at the site of vulvar biopsy will have lower pain scores on a visual analogue scale during the biopsy.

Study Design: Double blinded randomized controlled trial

Population: Women undergoing vulvar biopsy at the Women's Primary Care Center and The Program In Women's Oncology Clinic of a non-infectious vulvar lesion.

DETAILED DESCRIPTION:
BACKGROUND/INTRODUCTION:

Certain procedures, particularly those involving the skin, can cause pain and distress in patients. Often , a local anesthetic is used to dull the sensation and improve patient experience and satisfaction. The procedure at hand dictates the mode of delivery of the anesthetic, but typically immediate and fast acting analgesia requires infiltration. Lidocaine is in the amide class of local anesthetics and is the most commonly used agent for infiltration. Lidocaine is usually given as a 1 percent solution and can be combined with epinephrine in order to prolong the duration of action, decrease local bleeding via local vasoconstriction and decrease systemic absorption of the lidocaine.

It is well known that lidocaine injection can be painful, likely secondary to the acidity. A meta analysis published in the Cochrane Database of 23 trials that compared pain during infiltration of buffered or non-buffered lidocaine found that patients receiving buffered lidocaine reported significantly less pain than those who received non-buffered lidocaine. The decrease in pain was greater for patients who received lidocaine with epinephrine but was also present for those who received lidocaine without epinephrine. The authors' conclusion was that "increasing the pH of lidocaine decreased pain on injection and augmented patient comfort and satisfaction". The studies included in this review however were mainly focused on lacerations, carpal tunnel decompression and "outpatient procedures". There were two studies that specifically involved OB/GYN patients; one investigated buffered lidocaine during epidural catheter removal and the other investigated buffered lidocaine during Norplant insertion. Since the Cochrane Review was published, one further gynecologic study investigating buffered lidocaine has been published involving cervical loop excision.

To date, there are no studies investigating the efficacy of buffered lidocaine during procedures on the vulva. The vulva is a particularly sensitive region to have a biopsy performed because it has extensive innervation, a large blood supply and it involves a pelvic exam which can be associated with increased anxiety. As many OBGYNs know, the vulva can be affected by a variety of conditions both benign and malignant. A crucial aspect of caring for women with vulvar complaints is conducting biopsies of lesions to ensure no occult malignancy and/or to further classify a diagnosis with histology. Use of local anesthetic is standard of care during biopsy but can add to the pain and discomfort of an already painful procedure. Some sources recommend use of topical anesthetic prior to infiltration of lidocaine, particularly in the pediatric patient. However, this technique requires the topical anesthetic be applied 20-60 minutes prior to the biopsy, which may not be feasible in a busy outpatient practice. Currently, the American Board of Obstetrics and Gynecology suggests 8.4% sodium bicarbonate can be added to lidocaine to minimize discomfort. However, there is currently no standard anesthesia recommendations and this is often not being done in clinical practice.

Given the obstacles to topical anesthetic usage, the fact that it does not address the pain involved with lidocaine infiltration and the lack of published literature on use of buffered lidocaine on the vulva, this study aims to investigate the use of buffered lidocaine versus non-buffered lidocaine in the setting of vulvar biopsy using a visual analog scale.

Research Question: Does buffered lidocaine decrease pain scores on a visual analogue scale during infiltration for local anesthesia during vulvar biopsy?

METHODOLOGY/ STUDY DESIGN:

This study will be a double blinded, randomized controlled trial to be performed at the Women's Primary Care Center and The Program In Women's Oncology Clinics. Patients will be recruited as outlined below and assigned a sequential study identification number. They will be asked to complete the questions on the Data Collection Form/Survey (see form titled "Data Collection Form") and if they agree to the study, will sign the Informed Consent (see form titled "Informed Consent"). The Data Collection Form/Survey will be given to the patient upon decision to perform a vulvar biopsy by the provider. The patient will be consented by approved research personnel. Then, the patient will undergo a vulvar biopsy as per clinician protocol. Baseline pain scores will be collected using the visual analogue scale. After skin prep, the pre-filled, sequentially numbered, randomized 25 gauge syringes will be used to inject 3ml of either buffered or non-buffered lidocaine prepared by the pharmacy as outlined below. The biopsy will then proceed as per clinical standard. The patient will be presented a 100 mm visual analogue scale to mark their pain level. A total of three pain scores will be obtained as the patient marks on the pain scale when instructed: A baseline pain score prior to intervention, pain score at time of infiltration, and pain score at the completion of the biopsy. The Data Collection Form/Survey will be collected from the patient by approved research personnel and placed in secure storage. Data will be entered into a secure electronic database for statistical analysis. Nursing staff at the WPCC may be present for the biopsy, but will not be involved in the conduction of the study.

The study population of interest is patients undergoing vulvar biopsy for noninfectious lesions. These clinic sites were chosen for this project given the relatively high volume of such procedures. There are a number of other trials that have taken place or are ongoing at the Women's Primary Care Center and The Program In Women's Oncology Office, such that ample infrastructure and resources are available. Many of the patients have been approached for other research trials, and may be more willing to participate for that reason.

SAMPLE SIZE: The sample size calculation is based on the null hypothesis that the mean pain score will be the same in women treated with buffered lidocaine as in those treated with non-buffered placebo. The alternative hypothesis (two-sided) is that the mean pain score in women treated with buffered lidocaine will be different than those treated with non-buffered lidocaine. Assuming an alpha of 0.05, 80% power, and a standard deviation of 21-30 mm (based on a previous study measuring pain with tenaculum application and intracervical block), we will need to recruit 64 women per arm to be able to detect a 15 mm mean difference between groups on the 100 mm VAS. This difference is derived from a prior study showing the minimally clinically significant difference in acute pain on the VAS is 12 mm, with a 95% confidence interval range from 9 to 15 mm. Therefore, we plan to recruit a total of 128 patients, or 64 patients per arm.

CRITERIA FOR SUBJECT SELECTION/RECRUITMENT METHOD: Participants will be recruited from June 2015-April 2018. All patients at the Women's Primary Care Center and The Program In Women's Oncology Clinic who are to undergo a vulvar biopsy for a noninfectious vulvar lesion will be approached by the research assistant or provider in the clinic and asked to participate in the study. The research assistant/provider will then review the study protocol, risks, benefits, and the written informed consent form with the patient (see form titled "Informed Consent"). If the patient wishes to participate, written informed consent for the study will be obtained by study personnel prior to the biopsy. Women from all racial and ethnic groups will be considered for inclusion in this study and no person shall be excluded based on their race or ethnicity.

DATA COLLECTION/INTERPRETATION: All data will be collected prospectively by the research staff or nursing staff (nursing staff at the WPCC will not be involved in research activities). Before the biopsy, a questionnaire will be completed by the patient to identify any factors that may influence pain perceived during the biopsy as well as baseline demographic information: age, race/ethnicity, education level, any analgesics taken the day of the biopsy. The physician performing the biopsy and indication for the biopsy will also be noted. The primary outcome of interest will be pain score on the visual analogue scale during lidocaine infiltration. A total of three pain scores will be obtained by the research assistant or nurse: A baseline pain score prior to intervention, pain score at time of infiltration, and pain score at the completion of the biopsy. This will be measured by asking the patient to mark her pain level on a 100 mm scale at each predetermined time point.

The analysis plan is based on the primary outcome of mean pain score during lidocaine infiltration as measured on the 0 mm to 100 mm VAS. The investigators are comparing two groups: 1) buffered lidocaine 2) non-buffered lidocaine. If the data are normally distributed, we will compare mean pain scores between the two groups using a t-test. If the data deviate notably from normality, the nonparametric Wilcoxon rank sum test will be used for comparisons. Imbalances will be handled by adjustment for covariates in multiple linear regression. The investigators will use an intention to treat analysis.

After written informed consent is obtained and subjects are admitted into the study, participants will be randomized to one of two groups, buffered lidocaine or non-buffered lidocaine. Randomization lists will be computer generated with a one-to-one allocation ratio in blocks by the WIH pharmacy staff. After signing the consent form, each participant will be assigned a study ID number corresponding with the order of recruitment into the study. The pharmacy will prepare identical syringes containing 9 ml of the 1% lidocaine + 1 ml of sodium bicarbonate or 10 ml 1% lidocaine labeled only with the study name and sequentially numbered. The numbered syringe corresponding with the participant's study ID number will be obtained by the study staff from the locked refrigerator in the Women's Primary Care Center or The Program In Women's Oncology. The syringes will appear identical. Participants, study personnel, the medical assistant, and the clinician will be blinded to the assignment.

FACILITIES: All patient related aspects of the study will transpire in the Women's Primary Care Center and The Program In Women's Oncology. Data processing and interpretation will take place at Women and Infants Hospital in conjunction with the Division of Research.

CONFIDENTIALITY: The patients enrolled in the study will be asked permission for access to their medical records. To ensure patient confidentiality, all forms will be marked with only the participant ID number, with a key containing identifying information kept separately in a locked cabinet that only research personnel will have access to. Electronic data will be stored on the Care New England file server, a file server that is located in a physically secured data center. Access to Care New England data center is card-controlled and all access to the server room is recorded. Care New England computer account management policies and practices ensure that computer access to the study database will be limited to key study personnel.

SAFETY: Study personnel will meet to review safety issues and logistics at 25%, 50% and 75% recruitment. Adverse events and complications will be recorded on the data collection sheet which will be reviewed by the PI on a rolling basis.

PERSONNEL/ADMINISTRATION AND ORGANIZATIONAL STRUCTURE:

Patients will be recruited by and data collected by designated research staff and/or providers in the Women's Primary Care Center and The Program In Women's Oncology. The biopsies will be performed by designated key research personnel. These providers are educated on the standard protocol utilized by the Center. Nursing staff at the WPCC may be present for the biopsy, but will not be involved in the conduction of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the Women's Primary Care Center
* Ages 18 and older
* Require a vulvar biopsy for a noninfectious vulvar lesion.
* Able to read English or Spanish
* Able to give informed consent for involvement in the study

Exclusion Criteria:

* Allergy to lidocaine
* Unable to give informed consent
* Unable to read English or Spanish

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Pain scores on Visual Analogue Pain Scale (100mm) | Before procedure, approximately 5 minutes
Pain scores on Visual Analogue Pain Scale (100mm) | During infiltration of lidocaine, approximately 10 minutes
Pain scores on Visual Analogue Pain Scale (100mm) | After completion of procedure, approximately 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Villavicencio, MD, Principal Investigator — Women and Infants Hospital
Locations (2):
- United States (2):
  - Women and Infants Hospital, Program in Women's Oncology, Providence, Rhode Island
  - Women's Primary Care Center/Women and Infants' Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Villavicencio JC, Kulkarni A, Luis C, Mendez H, Raker C, Cronin B, Robison K. Sensation of Pain Using Buffered Lidocaine for Infiltration Before Vulvar Biopsy: A Randomized Controlled Trial. Obstet Gynecol. 2020 Mar;135(3):609-614. doi: 10.1097/AOG.0000000000003710. PMID 32028501